CLINICAL TRIAL: NCT07397026
Title: Clinical and Laboratory Evaluation of Resveratrol Loaded Nanoparticles in the Treatment of Periodontitis: A Randomized Controlled Clinical Trial
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hagar Ahmed Ali Mohammed Elzain (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Hagar Ahmed Ali Mohammed Elzain, clinical demonstrator faculty of dentistry Mansoura university, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M0102025OM
Record Dates: First submitted 2025-12-21; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Periodontitis Stage III
Keywords: Periodontitis; Resveratrol; Nanoparticles; Cox-2; Scaling; root planing; Gingival crevicular fluid; Superoxide dismutase
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (negative control group): includes 12 periodontally healthy subjects (No Intervention): Healthy Patients who are accepted for this study will be screened by a comprehensive periodontal examination and full periodontal charts. Proper Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017 AAP World Workshop.
  * Clinical periodontal parameters, including:
    1. Plaque Index (PI), according to Silness P. Loe H 1964.
    2. Gingival Index (GI), according to Silness P. Loe H 1963.
    3. Eastman Interdental Bleeding Index (EIBI), according to Ainamo & Bay 1975.
    4. Clinical Attachment Level (CAL) is measured from cemento enemal junction to base of the pocket.
    5. Probing Pocket Depth(PPD) is measured from free gingival margin to base of the pocket.
       ALL these parameters will be assessed at baseline.
  * GCF samples will be collected using sterile paper strips and analyzed using the commercially available kits for the assessment of the level of COX-2 and SOD at baseline .
  no injection of Resveratrol Loaded Nanoparticles .
- Group 2(positive control group): includes 12 patients will be treated with Scaling and root planing (Sham Comparator): Patients who are accepted for this study will be screened by periodontal examination and full periodontal charts. Proper Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017
  * Clinical periodontal parameters, including:
    1. Plaque Index (PI) .
    2. Gingival Index(GI) .
    3. Eastman Interdental Bleeding Index (EIBI) .
    4. Clinical Attachment Level (CAL) .
    5. Probing Pocket Depth(PPD) is measured from free gingival margin to base of the pocket.
       ALL these parameters will be assessed at baseline and after 3 months after treatment .
  * GCF samples will be collected using sterile paper strips and analyzed using the commercially available kits for the assessment of the level of COX-2 and SOD at baseline and after 3 months after treatment .
  After proper and accurate examination and diagnosis, full mouth supra- and subgingival SRP will be performed with ultrasonic tips and Gracey curettes .
  patients will receive oral hygiene instructions.
  Interventions: Drug: Resveratrol loaded gel
- Group 3 (placebo group): includes 12 patients will be treated with Resveratrol unloaded gel (Placebo Comparator): Patients who are accepted for this study will be screened by periodontal examination and full periodontal charts. Proper Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017
  * Clinical periodontal parameters, including:
    1. PI .
    2. GI .
    3. EIBI .
    4. CAL .
    5. PPD.
  * GCF samples will be collected using sterile paper strips and analyzed using the commercially available kits for the assessment of the level of COX-2 and SOD at baseline and after 3 months after treatment .
  After diagnosis, full mouth supra- and subgingival SRP will be performed with ultrasonic tips and Gracey curettes .
  patients will receive oral hygiene instructions.
  After completion of SRP, RES unloaded gel will be injected as placebo gel in using a syringe with a blunt cannula until the pocket will be completely filled.
  the Patients will be instructed to avoid chewing hard, eating any sticky foods for several hours.
  No intervention of Resveratrol Loaded Nanoparticles .
  Interventions: Drug: Resveratrol loaded gel
- Group 4 (Resveratrol Loaded Nanoparticles):12 patients will be injected with Resveratrol loaded gel (Other): Patients who are accepted for this study will be screened by periodontal examination and full periodontal charts. Proper Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017
  * Clinical periodontal parameters, including:
    1. PI .
    2. GI .
    3. EIBI .
    4. CAL .
    5. PPD.
  * GCF samples will be collected using sterile paper strips and analyzed using the commercially available kits for the assessment of the level of COX-2 and SOD at baseline and after 3 months after treatment .
  After diagnosis, full mouth supra- and subgingival SRP will be performed with ultrasonic tips and Gracey curettes .
  patients will receive oral hygiene instructions.
  After completion of SRP, Resveratrol loaded nanoparticles gel will be injected in the selected periodontal pocket using a syringe with a blunt cannula until the pocket will be completely filled.
  there is intervention by injection of Resveratrol Loaded Nanoparticles inside the pocket .
  Interventions: Drug: Resveratrol loaded gel

INTERVENTIONS:
Drug: Resveratrol loaded gel — Locally injection of Resveratrol Loaded Nanoparticles in patients with stage II periodontitis according to 2017 classification in group 4 only while group 3 will be injected with placebo also group 2 will be treated with only SRP but group 1 is the healthy group ,these participants will only be screened by a comprehensive periodontal examination and full periodontal charts. Proper Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017 AAP World Workshop and no intervention will be done .
  Other Names: (Resveratrol loaded gel ); Resveratrol Loaded Nanoparticles
  Arms: Group 2(positive control group): includes 12 patients will be treated with Scaling and root planing; Group 3 (placebo group): includes 12 patients will be treated with Resveratrol unloaded gel; Group 4 (Resveratrol Loaded Nanoparticles):12 patients will be injected with Resveratrol loaded gel

SUMMARY:
The Aim of this study is to test the effectiveness of locally applied resveratrol as an adjunct to scaling and root planing in the treatment of periodontitis (primary outcome) . Also to assess the level of COX-2 and superoxide dismutase (SOD) in the gingival crevicular fluid samples using the commercially available kits.

DETAILED DESCRIPTION:
Patients who are accepted for this study will be screened by a comprehensive periodontal examination and full periodontal charts. Proper Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017 AAP World Workshop.

* Clinical periodontal parameters, including:

  1. Plaque Index (PI), according to Silness P. Loe H 1964.
  2. Gingival Index (GI), according to Silness P. Loe H 1963.
  3. Eastman Interdental Bleeding Index (EIBI), according to Ainamo & Bay 1975 .
  4. Clinical Attachment Level (CAL) is measured from cemento enemal junction to base of the pocket.
  5. Probing Pocket Depth(PPD) is measured from free gingival margin to base of the pocket.

     ALL these parameters will be assessed at baseline and after 3 months after treatment for groups 2, 3 and 4 while at baseline only for group 1.
* GCF samples will be collected using sterile paper strips and analyzed using the commercially available kits for the assessment of the level of COX-2 and SOD at baseline and after 3 months after treatment for groups 2, 3 and 4 while at baseline only for group 1.

After proper and accurate examination and diagnosis, full mouth supra- and subgingival SRP will be performed with ultrasonic tips and Gracey curettes (Hu-Friedy, Chicago, United States) and an ultrasonic device (Minipiezon, EMS [Electro Medical System], Le Sentier, Switzerland). All patients will receive oral hygiene instructions. After completion of SRP, RES loaded gel will be injected in the selected periodontal pocket of the test group (group 4) while RES unloaded gel will be injected as placebo gel in group 3 using a syringe with a blunt cannula until the pocket will be completely filled.

After atraumatic application of the local drug delivery system, the Patients will be instructed to avoid chewing hard, eating any sticky foods for several hours.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient 25-55 years.
2. Presence of ≥20 teeth.
3. PPD >3&≤5 mm.
4. The patients are in good systemic health.
5. Patients have not received any periodontal surgery in the areas that will be assessed in the last 6 months

Exclusion Criteria:

1. Patients with systemic diseases.
2. Pregnant and lactating women.
3. Heavy Smokers and tobacco chewers.
4. Patients do not follow oral hygiene measures.
5. Patients with a known or suspected allergy to any material used in the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-08-09 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) as Clinical periodontal parameter | 3 months
  Patients who are accepted for this study will be screened by periodontal examination and full periodontal charts. Proper Diagnosis of the stages of periodontitis will be based on the new classification proposed in 2017.
  Clinical attachment level (CAL) as Clinical periodontal parameter in mm

SECONDARY OUTCOMES:
laboratory evaluation of Cox-2 & SOD in GCF | 3 months
  GCF samples will be collected using sterile paper strips and analyzed using the commercially available kits for the assessment of the level of COX-2 and SOD at baseline and after 3 months after treatment for groups 2, 3 and 4 while at baseline only for group 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry , Mansoura university, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kornman KS. Controlled-release local delivery antimicrobials in periodontics: Prospects for the future. Journal of periodontology. 1993;64:782-91.
- [Background] Goodson J, Haffajee A, Socransky S. Periodontal therapy by local delivery of tetracycline. Journal of Clinical Periodontology. 1979;6(2):83-92.
- [Background] Cobb CM. Clinical significance of non-surgical periodontal therapy: an evidence-based perspective of scaling and root planing. Journal of clinical periodontology. 2002;29:22-32.
- [Background] Page RC, Kornman KS. The pathogenesis of human periodontitis: an introduction. Periodontology 2000. 1997;14(1):9-11.
- [Background] Graves DT, Cochran D. The contribution of interleukin-1 and tumor necrosis factor to periodontal tissue destruction. Journal of periodontology. 2003;74(3):391-401.
- [Background] Darveau RP. Periodontitis: a polymicrobial disruption of host homeostasis. Nature reviews microbiology. 2010;8(7):481-90.
- [Background] Hajishengallis G. Periodontitis: from microbial immune subversion to systemic inflammation. Nature reviews immunology. 2015;15(1):30-44.
- [Background] 2. Socransky SS, Haffajee AD. Dental biofilms: difficult therapeutic targets. Periodontology 2000. 2002;28(1):12-55.
- [Background] 1. Hussein MH, Badr BM, Hassan KS, Ibrahim IH. Evaluation of the Effect of Topically Applied Resveratrol Gel as Adjunctive Treatment for Periodontitis. European Journal of General Dentistry. 2024.